CLINICAL TRIAL: NCT03215121
Title: Comparative Evaluation of One Handed Versus Two Handed Mask Holding Techniques in Children During Induction of Anesthesia
Brief Title: Mask Study: One-handed vs. Two Handed Technique in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Dinesh Choudhry, Pediatric Anesthesiologist and Director of Pain Service, Principal Investigator, Associate Professor of Anesthesiology, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1065828-2
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Childrenwith documented obstructive sleep apnea (by sleep study or history obtained from the parent) due to enlarged tonsils and adenoid scheduled for tonsillectomy and adenoidectomy surgery will be enrolled in the study. Children will be randomly divided in two groups of 20 each based on the induction technique used:
  Group --1: Induction of anesthesia started as follows while children are breathing spontaneously: One handed mask airway + chin lift - 20 sec and then switch to two hands + jaw thrust - 20 sec Group - 2: Induction of anesthesia started as follows while children are breathing spontaneously: Two handed mask airway + jaw thrust - 40 sec.
  Group 3 - Induction of anesthesia started as follows while children are breathing spontaneously. Two handed mask airway + jaw thrust - 20 sec. then switch to one hand + chin lift - 20 sec.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One handed mask airway, switch to two hands (Active Comparator): Induction of anesthesia started as follows while children are breathing spontaneously: One handed mask airway + chin lift - 20 sec and then switch to two hands + jaw thrust - 20 sec
  Interventions: Procedure: One handed mask airway, switch to two hands
- Two handed mask airway + jaw thrust (Active Comparator): Induction of anesthesia started as follows while children are breathing spontaneously: Two handed mask airway + jaw thrust - 40 sec
  Interventions: Procedure: Two handed mask airway + jaw thrust
- Two handed mask airway, switch to one hand (Active Comparator): Induction of anesthesia started as follows while children are breathing spontaneously: Two handed mask airway + jaw thrust - 20 sec and then switch to one hand + chin lift - 20 sec
  Interventions: Procedure: Two handed mask airway, switch to one hand

INTERVENTIONS:
Procedure: One handed mask airway, switch to two hands — Prior to the induction of anesthesia, a shoulder role will be used to have the child's head in sniffing position for induction. Horizontal alignment of the external auditory meatus with the sternum, will be used as a marker for, proper positioning.
  Oxygen and nitrous oxide for 10-15 seconds will be administered and sevoflurane will then be commenced.The provider will hold the mask as randomized, one hand mask airway with switch to two hand for Group 1 patients. Any changes in airway patency when mask is held by one hand versus two hands will be observed and documented by various parameters. The initial mask management will be performed for 20 seconds.
  After another 20 seconds (50 seconds from the start of induction), in Group one, the mask holding will switch to two hands for 20 seconds.
  Arms: One handed mask airway, switch to two hands
Procedure: Two handed mask airway + jaw thrust — Prior to the induction of anesthesia, a shoulder role will be used to have the child's head in sniffing position for induction. Horizontal alignment of the external auditory meatus with the sternum, will be used as a marker for, proper positioning.
  Oxygen and nitrous oxide for 10-15 seconds will be administered and sevoflurane will then be commenced.The provider will hold the mask as randomized, two hands for Group two patients. Any changes in airway patency when mask is held by one hand versus two hands will be observed and documented by various parameters. In Group 2 patient's mask will be held with two hands first for 40 seconds.
  Arms: Two handed mask airway + jaw thrust
Procedure: Two handed mask airway, switch to one hand — Prior to the induction of anesthesia, a shoulder role will be used to have the child's head in sniffing position for induction. Horizontal alignment of the external auditory meatus with the sternum, will be used as a marker for, proper positioning.
  Oxygen and nitrous oxide for 10-15 seconds will be administered and sevoflurane will then be commenced.The provider will hold the mask as randomized, two hands for Group 3 patients. Any changes in airway patency when mask is held by one hand versus two hands will be observed and documented by various parameters. The initial mask management will be performed for 20 seconds.
  After another 20 seconds (50 seconds from the start of induction), in Group 3, the mask holding will switch to one hand for 20 seconds.
  Arms: Two handed mask airway, switch to one hand

SUMMARY:
During induction of anesthesia in children, the investigators have observed significant variability in mask holding technique at our institution among different anesthesia practitioners. Some hold the face mask using one hand and others use two hands. The aim of our study is to comparatively evaluate the extent of airway obstruction in children whilst anesthetic mask is held with one hand with jaw thrust versus mask held using two hands with chin lift by anesthesia provider during induction of anesthesia in children.

DETAILED DESCRIPTION:
In a prospective, randomized and controlled study, 60 children with documented obstructive sleep apnea (from sleep study or history obtained from the parent of bothersome snoring, witnessed apnea which interrupts the snoring and/or gasping and choking sensations that arouse the patient from sleep) due to enlarged tonsils and adenoid scheduled for tonsillectomy and adenoidectomy surgery will be enrolled in the study. Children will be randomly divided in three groups of 20 each based on the induction technique used:

Group --1: Induction of anesthesia started as follows while children are breathing spontaneously: One handed mask airway + chin lift - 20 sec and then switch to two hands + jaw thrust - 20 sec

Group 2 - Induction of anesthesia started as follows while children are breathing spontaneously: Two handed mask airway + jaw thrust - 40 sec

Group 3 - Induction of anesthesia started as follows while children are breathing spontaneously: Two handed mask airway + jaw thrust - 20 sec and then switch to one hand + chin lift- 20 sec

Premedication with midazolam as per standard protocol, will be administered prior to taking the patients to the operating room. Prior to the induction of anesthesia, a shoulder role will be used to have the child's head in sniffing position for induction. Horizontal alignment of the external auditory meatus with the sternum, will be used as a marker for, proper positioning.

Oxygen and nitrous oxide for 10-15 seconds will be administered and sevoflurane will then be commenced. Addition of sevoflurane will be recorded as the start of induction. The provider will hold the mask as randomized, one hand with switch to two hands for Group 1 patients, two hands for Group 2 patients and two hands with switch to one hand for Group 3 patients. Any changes in airway patency when mask is held by one hand versus two hands will be observed and documented by various parameters stated below. The initial mask management will be performed for 20 seconds.

After another 20 seconds (50 seconds from the start of induction), mask holding will switch to two hands for 20 seconds. In Group 2 patients mask will be held with two hands for 40 seconds. No oropharyngeal or nasopharyngeal airway will be placed during the study period. In Group 3 patients, mask will initially be held with two hands for 20 seconds, with switch to one hand for 20 seconds.

In the investigators clinical experience, the rate of obstructive symptoms with one hand ventilation approaches 100% and obstructive symptoms with two hands ventilation approaches 0%. Using this ratio data for a power analysis to determine sample size yielded 4 subjects per group. As this is probably unreasonably low, the ratios were adjusted to 75% for one hand and 25% for two hand ventilation, which yielded 18 subjects per group to achieve an alpha of 95%, and beta of 80%. With the potential for case dropout, the sample sizes for this study were set at 20 per group to reasonably ensure statistical significance. Given that approximately 80 cases of tonsillectomy and adenoidectomy cases are performed due to obstruction a year, this sample size should be easily obtainable. Randomization of patient assignment to the groups will be accomplished by graph pad quickcalcs.

(http://www.graphpad.com/quickcalcs/randomize1.cfm).

Continuous variables, times and ratio data will be analyzed by t test and nominal data by chi square.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 to 8 years of age Scheduled for Tonsillectomy & adenoidectomy Documented evidence of obstructive sleep apnea ASA I and II

Exclusion Criteria:

* Children with abnormal airway anatomy ASA III and over

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Work of breathing | 20 - 40 seconds
  Phase angle

SECONDARY OUTCOMES:
Airway Obstruction Rating Scale 0 - 3 | 20-40 seconds
  Presence of airway obstruction:
  0= No obstruction; 1=Good gas exchange with noisy breathing, no retractions; 2=Mild retractions with diminished air flow; 3=Severe retractions with minimal/no air flow
Laryngospasm | 20-40 seconds
  Indicate presence: yes/no
Breath holding | 20-40 seconds
  Indicate presence: yes/no
Labored breathing | 20-40 seconds
  labored breathing index (RCI)
Rib cage movement | 20-40 seconds
  %Rib Cage movement (%RC)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours/A I duPont Hospital for Children, Wilmington, Delaware, United States

REFERENCES:
- [Background] Keidan I, Fine GF, Kagawa T, Schneck FX, Motoyama EK. Work of breathing during spontaneous ventilation in anesthetized children: a comparative study among the face mask, laryngeal mask airway and endotracheal tube. Anesth Analg. 2000 Dec;91(6):1381-8. doi: 10.1097/00000539-200012000-00014. PMID 11093984
- [Background] von Ungern-Sternberg BS, Erb TO, Reber A, Frei FJ. Opening the upper airway--airway maneuvers in pediatric anesthesia. Paediatr Anaesth. 2005 Mar;15(3):181-9. doi: 10.1111/j.1460-9592.2004.01534.x. No abstract available. PMID 15725313
- [Background] Litman RS, Kottra JA, Berkowitz RJ, Ward DS. Upper airway obstruction during midazolam/nitrous oxide sedation in children with enlarged tonsils. Pediatr Dent. 1998 Sep-Oct;20(5):318-20. PMID 9803430
- [Background] Rahman T, Page R, Page C, Bonnefoy JR, Cox T, Shaffer TH. pneuRIPTM: A Novel Respiratory Inductance Plethysmography Monitor. J Med Device. 2017 Mar;11(1):0110101-110106. doi: 10.1115/1.4035546. Epub 2017 Jan 24. PMID 28289485
- [Background] Kheterpal S. It's About Time. Anesthesiology. 2017 Jan;126(1):4-5. doi: 10.1097/ALN.0000000000001408. No abstract available. PMID 27811484
- [Background] Sato S, Hasegawa M, Okuyama M, Okazaki J, Kitamura Y, Sato Y, Ishikawa T, Sato Y, Isono S. Mask Ventilation during Induction of General Anesthesia: Influences of Obstructive Sleep Apnea. Anesthesiology. 2017 Jan;126(1):28-38. doi: 10.1097/ALN.0000000000001407. PMID 27811485
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Background] Kheterpal S, Han R, Tremper KK, Shanks A, Tait AR, O'Reilly M, Ludwig TA. Incidence and predictors of difficult and impossible mask ventilation. Anesthesiology. 2006 Nov;105(5):885-91. doi: 10.1097/00000542-200611000-00007. PMID 17065880
- [Background] Kheterpal S, Martin L, Shanks AM, Tremper KK. Prediction and outcomes of impossible mask ventilation: a review of 50,000 anesthetics. Anesthesiology. 2009 Apr;110(4):891-7. doi: 10.1097/ALN.0b013e31819b5b87. PMID 19293691